CLINICAL TRIAL: NCT02384668
Title: The DAGMAR Study. D-vitamin And Graves' Disease; Morbidity And Relapse Reduction: A Randomised, Clinical Trial.
Brief Title: D-vitamin And Graves' Disease; Morbidity And Relapse Reduction
Acronym: DAGMAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other); Regional Hospital Holstebro (Other); Regionshospitalet Horsens (Other); Randers Regional Hospital (Other); Regionshospitalet Viborg, Skive (Other); Herning Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12122012
Record Dates: First submitted 2015-01-09; First posted 2015-03-10 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Graves' Disease
Keywords: Cholecalciferol; Vitamin D3; Arterial stiffness; Quality of Life; Bone density and geometry; Muscle strength and balance
MeSH Terms: conditions — Graves Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Active Comparator): Cholecalciferol 70 mcg per day Other name: Vitamin D3.
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator): Placebo tablets are identical in regards to size and appearance to the experimental intervention tablet.
  The placebo regimen is identical to the vitamin D3 regimen.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — One tablet per day. The duration of the intervention period is between 24-36 months. This is defined by the time of ATD treatment withdrawal, which is scheduled between approximately 12-18(-24) months after randomisation. Vitamin D supplementation will continue 12 months after withdrawal of ATD treatment or until relapse of Graves' Disease if this occurs prior.
  Other Names: Vitamin D3
  Arms: Cholecalciferol
Dietary Supplement: Placebo — One tablet per day. Placebo tablet identical in appearance to cholecalciferol tablet. Duration and cessation of treatment identical to intervention with cholecalciferol.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of vitamin D supplementation on morbidity and risk of relapse in patients with Graves' disease.

DETAILED DESCRIPTION:
In a multicentre trial, 260 patients with newly diagnosed Graves ' disease will be randomized to cholecalciferol 70 mcg/day or placebo in a parallel Group design. Drop outs prior to 31th of December 2017 will be replaced. The intervention will continue during treatment with antithyroid drugs (ATD), and for a period of 12 months after cessation of ATD. Blood samples will be collected at study entry, at 3 and 9 months, and at end of study. QoL questionnaires on nine occasions through out the study period. In a subcohort of 80 participants detailed examinations of bone density and geometry, muscle strength and postural balance, immune tests (N=50), and measurements of arterial stiffness will be performed at study entry, and at 3 and 9 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* A first time diagnosis of Graves' hyperthyroidism within the last three months, confirmed by TSH below 0.01 IU/L, and T3 or T4 levels above the reference interval necessitating ATD therapy
* Positive TRAb
* Speak and read Danish
* Written informed consent

Exclusion Criteria:

* Previously diagnosed hyperthyroidism
* ATD treatment initiated more than 3 months prior to inclusion
* Planned ablative therapy (radioactive iodine or thyroid surgery)
* Intake of more than 10 µg D-vitamin/day that the participant wishes to continue.
* Chronic granulomatous illness
* Persistent hypercalcemia (plasma calcium > 1.40 mmol/L)
* Reduced kidney function (eGFR < 45 ml/min)
* Treatment with immunomodulatory drugs
* Active malignant disease
* Alcohol or drug abuse
* Pregnancy at inclusion
* Major comorbidity, making the participant unlikely to continuously receive trial intervention.
* Allergy towards the components in the D-vitamin or the placebo pills.
* Unable to read and understand Danish
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants without relapse within the first year after cessation of ATD treatment. | 0-12 months after cessation of ATD treatment
  A relapse is defined as:
  The participant has been referred to radioactive iodine or thyroid surgery at any time during the entire intervention period; or The participant has hyperthyroidism (TSH<0.1) at 12 months (+/- 1 months) after cessation of ATD treatment; or ATD is re-initiated within 12 months after cessation of initial ATD treatment; or The participant fails to stop ATD treatment within 24 months after initiation of ATD treatment.

SECONDARY OUTCOMES:
The proportion of participants who has been referred to radioactive iodine or thyroid surgery at any time during the entire intervention period. | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  The proportion of participants who has been referred to radioactive iodine or thyroid surgery at any time during the entire intervention period.
The proportion of participants who have relapse of hyperthyroidism (TSH<0.1) after cessation of ATD therapy | 0-12 months after cessation of ATD treatment
  The proportion of participants who have relapse of hyperthyroidism (TSH<0.1) after cessation of ATD therapy
The proportion of participants who re-initiates ATD treatment or is referred to radioactive iodine or thyroid surgery due to hyperthyroidism within 12 months after cessation of initial ATD treatment. | 0-12 months after cessation of ATD treatment
  The proportion of participants who re-initiates ATD treatment or is referred to radioactive iodine or thyroid surgery due to hyperthyroidism within 12 months after cessation of initial ATD treatment.
The proportion of participants who fails to stop ATD treatment within 24 months after initiation of ATD therapy. | 0-24 months after initiation of ATD therapy
  In a pre-planned sub-analysis participants on sustained ATD treatment for more than 24 months after initiation of ATD therapy because of Graves' orbitopathy will be excluded
Effects of D-vitamin supplementation according to plasma level of D-vitamin at inclusion to the study. | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Sub analysis of all primary and secondary outcome measures will be performed according to this criteria.
Proportion of participants without relapse within the first year after cessation of ATD treatment according to baseline use of D-vitamin. | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Sub analysis of baseline "users" versus "non-users" of D-vitamin supplementation with regards to effects of intervention on all primary and secondary outcome measures.
Quality of Life as measured by Health questionnaires | 6 weeks
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Quality of Life as measured by Health questionnaires | 3 months
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Quality of Life as measured by Health questionnaires | 6 months
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Quality of Life as measured by Health questionnaires | 9 months
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Quality of Life as measured by Health questionnaires | 12 months
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Quality of Life as measured by Health questionnaires | 18 months
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Quality of Life as measured by Health questionnaires | 24 months
  Thyroid specific QoL as measured by the global score in the thyPRO questionnaire.
  Hyperthyroid symptoms (thyPRO subscale) Proportion of patients with eye symptoms (thyPRO subscale)
Biomarkers of calcium- and bone metabolism. | 3 months, 9 months and 12 months after cessation of ATD treatment, an expected average of 24 months
  Effects of intervention on biochemical markers of calcium and bone metabolism, such as calcium, phosphate, parathyroid hormone, calcitriol, vitamin D-binding protein, bone-specific alkaline phosphatase, osteocalcin, and N-terminal propeptide of type 1 procollagen (P1NP). Also C-terminal telopeptide of type 1 collagen (CTX) and N-telopeptide of type 1 collagen (NTX) among others.
Level of Thyrotropin receptor antibody (TRAb) | 3 months, 9 months and 12 months after cessation of ATD treatment, an expected average of 24 months
  Level of TRAb at 3 and 9 months and at end of study period (maximum of 36 months)
Level of 25 hydroxy vitamin D | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Level of 25 hydroxy vitamin D at 3 and 9 months and at end of study period (maximum of 36 months)

OTHER OUTCOMES:
Immune response as measured by flow cytometric analysis of T- and B-cells | First nine months.
  In a subcohort of 50 participants blood samples will be investigated by flow cytometry. Lymphocyte subpopulations will be quantified.
Immune response as measured by soluble HLA-G (Human Leukocyte Antigen-G) | First nine months.
  In a subcohort of 50 participants soluble HLA-G (Human Leukocyte Antigen-G) will be quantified based on blood samples.
Immune response as measured by membrane-bound HLA-G (Human Leukocyte Antigen-G) | First nine months.
  In a subcohort of 50 participants membrane-bound HLA-G (Human Leukocyte Antigen-G) will be quantified based on expression on monocytes.
Immune response assessed by qualitative analysis of regulatory T lymphocytes | First nine months.
  In a subcohort of 50 participants functional analysis of the suppressive capacity of regulatory T lymphocytes will be measured at 3 and 9 months after randomisation.
Arterial stiffness as measured by tonometry | First nine months
  Indices of arterial stiffness at 3 and 9 months after randomisation in a subcohort of 80 participants
Muscle strength and balance as measured by isometric tests and dynamic stability tests. | First nine months
  Effects on muscle strength (isometric tests of flexion and extension of thigh and hand), two function-tests (timed up-and go and timed stand-and-sit), and postural stability at 3 and 9 months after randomisation in a subcohort of 80 participants
Bone density and geometry as measured by DXA and HRpQCT scans | First nine months
  Bone density, geometry, and quality as assessed by dual energy x-ray absorptiometry (DXA) and high resolution peripheral quantitative computed tomography (HRpQCT)-scans 9 months months after randomisation in a subcohort of 80 participants
Effect on thyroid gland size by ultrasound examination | First nine months
  Estimation of thyroid volume by ultrasound examination
Proportion of patients with adverse reactions to anti thyroid drugs | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Proportion of patients with adverse reactions to anti thyroid drugs measured by regular questionnaires and reported complaints and events in patient journals
Proportion of patients with serious adverse events | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Based on reports from patients journals and hospitals admissions of agranulocytosis, leukopenia, aplastic anemia, hepatitis, and vasculitis
Effects on frequency of infectious disease as measured by use of antibiotics | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Data from the Danish prescription database
Effects on use of Health care services as measured by hospital admissions and visits to general practitioner | From randomisation until 12 months after cessation of ATD treatment, an expected average of 24 months
  Measured by all cause-hospital admissions and visits to general practitioner

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, Professor, Principal Investigator — Aarhus University Hospital
Locations (8):
- Denmark (8):
  - Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus C
  - Gentofte Hospital, Gentofte Municipality
  - Department of Internal Medicine, Regionshospitalet Herning, Herning
  - Department of Internal Medicine, Regionshospitalet Holstebro, Holstebro
  - Department of Internal Medicine, Regionshospitalet Horsens, Horsens
  - Department of Internal Medicine, Regionhospitalet Randers, Randers
  - Department of Internal Medicine, Diagnostisk Center, Regionshospitalet Silkeborg, Silkeborg
  - Department of Internal Medicine, Regionshospitalet Viborg, Viborg

REFERENCES:
- [Derived] Grove-Laugesen D, Ebbehoj E, Watt T, Hansen KW, Rejnmark L. Changes in bone density and microarchitecture following treatment of Graves' disease and the effects of vitamin D supplementation. A randomized clinical trial. Osteoporos Int. 2024 Dec;35(12):2153-2164. doi: 10.1007/s00198-024-07241-y. Epub 2024 Sep 12. PMID 39264438
- [Derived] Grove-Laugesen D, Ebbehoj E, Watt T, Riis AL, Ostergard T, Bruun BJ, Juel Christiansen J, Hansen KW, Rejnmark L. Effect of Vitamin D Supplementation on Graves' Disease: The DAGMAR Trial. Thyroid. 2023 Sep;33(9):1110-1118. doi: 10.1089/thy.2023.0111. Epub 2023 Jun 26. PMID 37218433
- [Derived] Bislev LS, Wamberg L, Rolighed L, Grove-Laugesen D, Rejnmark L. Effect of Daily Vitamin D3 Supplementation on Muscle Health: An Individual Participant Meta-analysis. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1317-1327. doi: 10.1210/clinem/dgac004. PMID 35018442
- [Derived] Grove-Laugesen D, Cramon PK, Malmstroem S, Ebbehoj E, Watt T, Hansen KW, Rejnmark L. Effects of Supplemental Vitamin D on Muscle Performance and Quality of Life in Graves' Disease: A Randomized Clinical Trial. Thyroid. 2020 May;30(5):661-671. doi: 10.1089/thy.2019.0634. Epub 2020 Feb 7. PMID 31910101
- [Derived] Grove-Laugesen D, Malmstroem S, Ebbehoj E, Riis AL, Watt T, Hansen KW, Rejnmark L. Effect of 9 months of vitamin D supplementation on arterial stiffness and blood pressure in Graves' disease: a randomized clinical trial. Endocrine. 2019 Nov;66(2):386-397. doi: 10.1007/s12020-019-01997-8. Epub 2019 Jul 6. PMID 31280470

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT02384668/Prot_SAP_000.pdf
  • Informed Consent Form (2013-01-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT02384668/ICF_001.pdf